CLINICAL TRIAL: NCT00328926
Title: A Phase IV, Multicenter, Randomized, Double-blinded, Clinical Trial to Confirm the Efficacy of the 75 IU Dose of Luveris® vs. Placebo When Administered With Follitropin Alfa for Induction of Follicular Development and Pregnancy in Hypogonadotropic Hypogonadal Women With Profound LH Deficiency, as Defined by a Baseline LH Level <1.2 IU/L
Brief Title: Luveris® (Lutropin Alfa for Injection) in Women With Hypogonadotropic Hypogonadism (Luteinizing Hormone [LH] Less Than [<] 1.2 International Unit Per Liter [IU/L])
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Please see "Purpose" statement
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26109
Record Dates: First submitted 2006-05-20; First posted 2006-05-24 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: Hypogonadotropic Hypogonadism (LH <1.2 IU/L); Placebo; Luveris® 75 IU; Luveris® 25 IU; Recombinant human chorionic gonadotropin (r-hCG)
MeSH Terms: conditions — Hypogonadism | interventions — Luteinizing Hormone, beta Subunit; Glycoprotein Hormones, alpha Subunit; follitropin alfa; Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Luveris® 75 IU (Active Comparator)
  Interventions: Drug: Luveris® 75 IU; Drug: Recombinant human follicle stimulating hormone (r-hFSH); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- Luveris® 25 IU (Active Comparator)
  Interventions: Drug: Luveris® 25 IU; Drug: Recombinant human follicle stimulating hormone (r-hFSH); Drug: Recombinant human chorionic gonadotropin (r-hCG)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Recombinant human follicle stimulating hormone (r-hFSH); Drug: Recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: Luveris® 75 IU — Recombinant human luteinizing hormone (r-hLH, lutropin alfa, Luveris®), 75 IU will be administered subcutaneously once daily. Duration of treatment cycle will be up to 14 days, or maximum of 21 days (if follicular maturation is imminent, based upon follicular growth and estradiol [E2] levels). Total duration will be of 3 treatment cycles.
  Other Names: Lutropin alfa; Recombinant human luteinizing hormone (r-hLH)
  Arms: Luveris® 75 IU
Drug: Luveris® 25 IU — Recombinant human luteinizing hormone (r-hLH, lutropin alfa, Luveris®), 25 IU will be administered subcutaneously once daily. Duration of treatment cycle will be up to 14 days, or maximum of 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration will be of 3 treatment cycles.
  Other Names: Lutropin alfa; Recombinant human luteinizing hormone (r-hLH)
  Arms: Luveris® 25 IU
Drug: Placebo — Placebo will be administered subcutaneously once daily. Duration of treatment cycle will be up to 14 days, or maximum of 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration will be of 3 treatment cycles.
  Arms: Placebo
Drug: Recombinant human follicle stimulating hormone (r-hFSH) — Fixed dose of recombinant human follicle stimulating hormone (r-hFSH, follitropin alfa) 75 to 150 IU will be administered subcutaneously for 7 days. After 7 days of treatment, if the subject response will suboptimal, based on follicular growth and serum E2 levels, follitropin alfa dose adjusted to maximal dose of 225 IU. Duration of treatment cycle will be up to 14 days, or maximum of 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration will be of 3 treatment cycles.
  Other Names: Follitropin alfa
Drug: Recombinant human chorionic gonadotropin (r-hCG) — When the follicular response will adequate, ovulation will be triggered by a single 250 microgram subcutaneous injection of recombinant human chorionic gonadotropin (r-hCG, choriogonadotropin alfa). Duration of treatment cycle will be up to 14 days, or maximum of 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration will be of 3 treatment cycles.
  Other Names: Choriogonadotropin alfa

SUMMARY:
Sponsor has decided to discontinue Luveris® in the United States (US) due to level of customer demand for this product, and not due to any efficacy or safety concerns.

DETAILED DESCRIPTION:
To confirm the efficacy of the 75 IU dose of Luveris® compared to placebo when administered concomitantly with follitropin alfa for induction of clinical pregnancy in women with hypogonadotropic hypogonadism and profound LH deficiency (LH <1.2 IU/L), and to study the efficacy of a lower dose (25 IU) of Luveris® compared to placebo when administered concomitantly with follitropin alfa for induction of follicular development in women with hypogonadotropic hypogonadism and profound LH deficiency (LH <1.2 IU/L).

ELIGIBILITY:
Inclusion Criteria:

* Be premenopausal, between 18 and 40 years of age inclusive on the day of consent
* Have a clinical history of hypogonadotropic hypogonadism (World health organization [WHO] Group I type of anovulation) on the basis of congenital or acquired hypothalamic or pituitary endocrine dysfunction in the presence of qualifying screening laboratories
* Have no prior treatment cycles with gonadotropins or gonadotropin releasing hormone (GnRH) (gonadotropin naïve)
* Have discontinued estrogen-progesterone replacement therapy at least one month before the screening procedure
* Have primary or secondary amenorrhea
* Have a negative progestin challenge test performed during Screening
* Have the following hormonal values in a centrally analyzed fasting blood sample, drawn within 6 weeks before initiation of treatment:

  * Follicle-Stimulating Hormone (FSH): less than (<)5 international unit per liter (IU/L)
  * Leutinizing hormone (LH): <1.2 IU/L (a second Baseline serum LH level will be repeated two weeks after the initial LH draw)
  * Prolactin: < 43.3 nanogram per milliliter (ng/mL) (<1040 milli-international unit per liter [mIU/L])
  * Thyroid Stimulating Hormone (TSH): <6.5 micro-international units per milliliter (mcIU/mL)
  * Free Thyroxin (T4): 0.8-1.8 nanogram per deciliter (ng/dL) (11-24 picomole per liter [pmol/L])
  * Testosterone: <1.0 ng/mL (<3.5 nanomole per liter [nmol/L])
* Have an endovaginal pelvic ultrasound scan showing (i) no clinically significant uterine abnormality, (ii) no ovarian tumor or cyst, and (iii) less than or equal to (=<)13 small follicles (mean diameter =<10 milliliter [mm]) on the largest section through each ovary
* Have a normal cervical pap smear within 6 months of the initial visit
* Where indicated, have a normal or unchanged computed tomography (CT) scan or nuclear magnetic resonance (NMR) scan of the hypothalamic pituitary region on file
* Have a body mass index (BMI) between 18.4 and 31.4 kilogram per square meter (kg/m^2)
* Be willing and able to comply with the protocol for the duration of the study
* Have given written informed consent prior to any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to her future medical care

Exclusion Criteria:

* Any medical condition which in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug
* Any pre-existing medical condition which would compromise the subject's ability to conceive in vivo or to successfully complete a pregnancy
* Ongoing pregnancy
* Clinically important systemic disease (example: insulin-dependent diabetes mellitus, epilepsy, serious migraine, intermittent purpura, hepatic, renal or cardiovascular disease, serious corticoid-dependent asthma)
* Known infection with human immunodeficiency virus (HIV), Hepatitis B or C
* Ovarian enlargement or cyst of unknown etiology
* Abnormal gynecological bleeding of undetermined origin
* Previous or current hormone dependent tumor
* Known active substance abuse or eating disorder
* Known central nervous system (CNS) Lesions: In cases where hypogonadotropic hypogonadism (HH) is secondary to a CNS lesion or its treatment
* Exercise program exceeding 10 hours per week
* Is planning to undergo in vitro fertilization, intracytoplasmic sperm injection or another assisted reproductive technology (ART) procedure, other than intrauterine insemination, in the course of a study treatment cycle
* Currently undergoing treatment with psychotropic medication or with any other medication known to interfere with normal reproductive function (example: neuroleptics, dopamine antagonists)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono S.A., Geneva
Locations (1):
- U.S. Medical Information, 1-888-275-7376, Rockland, Massachusetts, United States

REFERENCES:
- See also: Full FDA approved prescribing information can be found here — http://fertilitylifelines.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Luveris® 75 IU: Recombinant human luteinizing hormone (r-hLH, lutropin alfa, Luveris®), 75 international unit (IU) administered subcutaneously once daily along with fixed dose of recombinant human follicle stimulating hormone (r-hFSH, follitropin alfa) 75 to 150 IU subcutaneously for 7 days. After 7 days of treatment, if the participant's response was suboptimal, based on follicular growth and serum estradiol (E2) levels, follitropin alfa dose adjusted to maximal dose of 225 IU. When the follicular response was adequate, ovulation was triggered by a single 250 microgram subcutaneous injection of recombinant human chorionic gonadotropin (r-hCG, choriogonadotropin alfa). Duration of treatment cycle was up to 14 days, or maximum up to 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration was up to 3 treatment cycles.
- Luveris® 25 IU: Recombinant human luteinizing hormone (r-hLH, lutropin alfa, Luveris®), 25 IU administered subcutaneously once daily along with fixed dose of recombinant human follicle stimulating hormone (r-hFSH, follitropin alfa) 75 to 150 IU subcutaneously for 7 days. After 7 days of treatment, if the participant's response was suboptimal, based on follicular growth and serum E2 levels, follitropin alfa dose adjusted to maximal dose of 225 IU. When the follicular response was adequate, ovulation was triggered by a single 250 microgram subcutaneous injection of recombinant human chorionic gonadotropin (r-hCG, choriogonadotropin alfa). Duration of treatment cycle was up to 14 days, or maximum up to 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration was up to 3 treatment cycles.
- Placebo: Placebo administered subcutaneously once daily along with fixed dose of recombinant human follicle stimulating hormone (r-hFSH, follitropin alfa) 75 to 150 IU subcutaneously for 7 days. After 7 days of treatment, if the participant's response was suboptimal, based on follicular growth and serum E2 levels, follitropin alfa dose adjusted to maximal dose of 225 IU. When the follicular response was adequate, ovulation was triggered by a single 250 microgram subcutaneous injection of recombinant human chorionic gonadotropin (r-hCG, choriogonadotropin alfa). Duration of treatment cycle was up to 14 days, or maximum up to 21 days (if follicular maturation is imminent, based upon follicular growth and E2 levels). Total duration was up to 3 treatment cycles.
Period: Overall Study
Arm/Group | Luveris® 75 IU | Luveris® 25 IU | Placebo
Started | 5 | 3 | 3
Completed | 3 | 0 | 1
Not Completed | 2 | 3 | 2
Not completed — Pregnancy | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1
Not completed — In vitro fertilization treatment | 0 | 0 | 1
Not completed — Lack of ovarian response | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luveris® 75 IU | Luveris® 25 IU | Placebo | Total
Number analyzed (Participants) | 5 | 3 | 3 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 28.6 (2.5) | 34.3 (5.0) | 29.3 (3.8) | 30.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 11
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Pregnancy
Description: Clinical pregnancy was defined as the presence of one or more fetal sac with fetal heart activity on the Day 35-42 post r-hCG ultrasound examination.
Time Frame: Stimulation Day 1 up to clinical pregnancy (Day 35-42 post r-hCG administration day [end of stimulation cycle {approximately 21 days}])
Population: Intention-to-treat (ITT) population included all the participants who received study treatment. 'N' (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Luveris® 75 IU | Luveris® 25 IU | Placebo
Number analyzed (Participants) | 3 | 1 | 1
Days | 71 [47 to 116] | 51 [51 to 51] | 103 [103 to 103]

2. Secondary Outcome: Percentage of Participants With Cumulative Clinical Pregnancy
Description: Clinical pregnancy was defined as the presence of one or more fetal sac with fetal heart activity on the Day 35-42 post r-hCG ultrasound examination. Cumulative clinical pregnancy referred to all clinical pregnancy that occurred during all the 3 treatment cycles.
Time Frame: Day 35-42 post r-hCG administration day (end of stimulation cycle [approximately 21 days])
Population: ITT population included all the participants who received study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Luveris® 75 IU | Luveris® 25 IU | Placebo
Number analyzed (Participants) | 5 | 3 | 3
Percentage of participants | 60.0 | 33.3 | 33.3

3. Secondary Outcome: Percentage of Participants With Cumulative Ovulation
Description: Ovulation was defined as a mid-luteal phase progesterone (P4) level greater than or equal to (>=) 10 nanogram per milliliter (ng/mL). Cumulative ovulation referred to all ovulations that occurred during all the 3 treatment cycles.
Time Frame: Recombinant human chorionic gonadotropin (r-hCG) administration day (end of stimulation cycle [approximately 21 days])
Population: ITT population included all participants who were treated to trial treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Luveris® 75 IU | Luveris® 25 IU | Placebo
Number analyzed (Participants) | 5 | 3 | 3
Percentage of participants | 80.0 | 33.3 | 66.7

ADVERSE EVENTS:
Time Frame: Stimulation Day 1 up to Day 35-42 post r-hCG administration day (end of stimulation cycle [approximately 21 days])
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an investigational medicinal product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Luveris® 75 IU | Luveris® 25 IU | Placebo
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 4/5 | 1/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luveris® 75 IU (N=5) | Luveris® 25 IU (N=3) | Placebo (N=3)
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luveris® 75 IU (N=5) | Luveris® 25 IU (N=3) | Placebo (N=3)
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysstasia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 1
Irritability (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Adnexa uteri pain (Reproductive system and breast disorders) | 3 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 2 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovulation pain (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other